CLINICAL TRIAL: NCT01323530
Title: A Phase 1b/2, Multicenter, Open-Label, Dose-Escalation and Confirmation Study of Eribulin in Combination With Capecitabine
Brief Title: A Confirmation Study of Eribulin in Combination With Capecitabine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: E7389-E044-203; 2009-011217-24 (EudraCT Number)
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-08

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose-escalation Phase (Phase 1b) (Experimental): Participants with advanced and/or metastatic tumors will receive eribulin mesylate as a 2 to 5 min Intravenous (IV) bolus or infusion in two different schedules (Schedule 1 [1.2, 1.6, 2.0 mg/m2], given on Day 1 only, and Schedule 2 [0.7, 1.1, 1.7 mg/m^2], given on Days 1 and 8) and oral capecitabine 1000 mg/m2 bid on Days 1-14 (21-day cycles) in both schedules. If maximum tolerated dose (MTD) is not observed at dose level 3 the dose of capecitabine might be escalated to 1250 mg/m^2 bid on Days 1-14 (21-day cycles) depending on the Dose limiting toxicities (DLTs) observed and/or pharmacokinetic (PK) data when available. Based on the data and safety monitoring board review of dose escalation phase data (DLTs that will be observed in first cycle), Dose-Confirmation Phase (Phase 2) will may get initiated.
  Interventions: Drug: Eribulin mesylate; Drug: Capecitabine
- Dose-confirmation Phase (Phase 2) (Experimental): Participants with advanced and/or metastatic tumors will receive Eribulin mesylate at the MTD for the selected schedule of dose escalation phase based on safety/PK data.
  Interventions: Drug: Eribulin mesylate; Drug: Capecitabine

INTERVENTIONS:
Drug: Eribulin mesylate — Intravenous (IV) bolus or infusion.
Drug: Capecitabine — Oral film-coated tablets.

SUMMARY:
This is a Phase 1b/2, multi-center, open-label, dose escalation (in 2 different dosing schedules [1 and 2]) and dose-confirmation study of eribulin administered in combination with capecitabine.

ELIGIBILITY:
Inclusion Criteria

Subjects who meet all of the following criteria will be included in the study:

Dose-escalation cohorts (Phase 1b):

1. Histologically or cytologically confirmed cancer that is advanced and/or metastatic
2. Resistant/refractory to approved therapies (defined as progressive disease during or within 6 months after the last anti-cancer therapy) or for whom single agent capecitabine at this dose level and schedule would be a reasonable treatment option in the opinion of the investigator
3. For subjects that previously received capecitabine, all capecitabine related toxicities must have completely resolved
4. Adequate bone marrow function as evidenced by absolute neutrophil count (ANC) greater than or equal to 1.5 x 10^9/L, hemoglobin greater than or equal to 10.0 g/dL (this may have been corrected by growth factor or transfusion), and platelet count greater than or equal to 100 x 10^9/L
5. Adequate liver function as evidenced by bilirubin less than or equal to 1.5 times the upper limit of normal (ULN) and alkaline phosphatase (AP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 x ULN (in the case of liver metastases less than or equal to 5 x ULN). In case AP is greater than 3 x ULN (in absence of liver metastases) or greater than 5 x ULN (in presence of liver metastases) AND subject also is known to have bone metastases, the liver specific AP must be separated from the total and used to assess the liver function instead of the total AP.
6. Adequate renal function as evidenced by calculated creatinine clearance greater than or equal to 50 mL/min as per the Cockcroft-Gault formula (Appendix 1) or radioisotope measurement.
7. Females of childbearing potential must have a negative urine or serum beta human chorionic gonadotropin (hCG) at Visit 1 (Screening) and prior to starting study drugs on Day 1. Female subjects of childbearing potential must agree to be abstinent or to use highly effective methods of contraception (e.g., condom + spermicide, condom + diaphragm with spermicide, intrauterine device (IUD), or have a vasectomized partner) having starting for at least one menstrual cycle prior to starting study drug(s) and throughout the entire study period and for 30 days (longer if appropriate) after the last dose of study drug. Those women using hormonal contraceptives must also be using an additional approved method of contraception (as described previously). Perimenopausal women must be amenorrheic for at least 12 months to be considered of nonchildbearing potential.
8. Male subjects who are not abstinent or have not undergone a successful vasectomy, who are partners of women of childbearing potential must use, or their partners must use, a highly affective method of contraception (e.g. condom + spermicide, condom + diaphragm with spermicide, IUD) starting for at least one menstrual cycle prior to starting study drug(s) and throughout the entire study period and for 30 days (longer if appropriate) after the last dose of study drug. Those with partners using hormonal contraceptives must also be using an additional approved method of contraception (as described previously)
9. Life expectancy of greater than 3 months
10. Willing and able to comply with all aspects of the protocol
11. Provide written informed consent
12. Eastern Cooperative Oncology Group (ECOG) performance status (PS) less than or equal to 2
13. Males and females, age greater than or equal to18 years

Dose-confirmation cohorts (Phase 2):

1. Histologically or cytologically confirmed carcinoma of the breast that is advanced and/or metastatic
2. Received up to three prior chemotherapy regimens in any setting (sequential neoadjuvant/ adjuvant treatment counting as one regimen)
3. Chemotherapy regimens must have included an anthracycline (unless anthracycline containing chemotherapy is inappropriate) and a taxane, either in combination or in separate regimens
4. No prior treatment with capecitabine in any setting
5. At least one lesion of greater than or equal to 1.5cm in longest diameter for non-lymph nodes and greater than or equal to 1.5cm in shortest diameter for lymph nodes which is serially measurable according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 7
6. Adequate bone marrow function as evidenced by ANC greater than or equal to 1.5 x 10^9/L, hemoglobin greater than or equal to 10.0 g/dL (this may have been corrected by growth factor or transfusion), and platelet count greater than or equal to 100 x 10^9/L
7. Adequate liver function as evidenced by bilirubin less than or equal to 1.5 times the upper limits of normal (ULN) and alkaline phosphatase (AP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal 3 x ULN (in the case of liver metastases less than or equal to 5 x ULN). In case AP is greater than 3 x ULN (in absence of liver metastases) or greater than 5 x ULN (in presence of liver metastases) AND subject also is known to have bone metastases, the liver specific AP must be separated from the total and used to assess the liver function instead of the total AP.
8. Adequate renal function as evidenced by calculated creatinine clearance greater than or equal to 50 mL/min as per the Cockcroft-Gault formula (Appendix 1) or radioisotope measurement.
9. Females of childbearing potential must have a negative urine or serum beta hCG at Visit 1 (Screening) and prior to starting study drugs on Day 1. Female subjects of childbearing potential must agree to be abstinent or to use highly effective methods of contraception (e.g., condom + spermicide, condom + diaphragm with spermicide, IUD, or have a vasectomized partner) having starting for at least one menstrual cycle prior to starting study drug(s) and throughout the entire study period and for 30 days (longer if appropriate) after the last dose of study drug. Those women using hormonal contraceptives must also be using an additional approved method of contraception (as described previously). Perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential
10. Life expectancy of greater than 3 months
11. Willing and able to comply with all aspects of the protocol
12. ECOG-PS 0 or 1
13. Females, age greater than or equal to 18 years

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from participation in the study:

1. Radiotherapy, chemotherapy, biological therapy or investigational agents within 4 weeks prior to the start of study treatment; subjects must have recovered from any previous therapy related toxicity to less than Grade 1 at study entry (except for stable sensory neuropathy less than or equal to Grade 2 and alopecia)
2. Treatment with mitomycin C or nitrosourea within 6 weeks prior to commencing on study treatment
3. Hormonal treatment within 2 weeks prior to start of study treatment (continued use of antiandrogens and/or gonadorelin analogues for treatment of prostate cancer permitted)
4. Prior participation in an eribulin clinical study, even if not assigned to eribulin treatment
5. Subject with hypersensitivity to halochondrin B and /or halochondrin B chemical derivates or capecitabine or any of the excipients
6. Suspected dihydropyrimidine dehydrogenase (DPD) deficiency
7. Previous radiotherapy encompassing greater than 30% of marrow
8. Previous organ allograft requiring immunosuppression
9. Subjects with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication at least 4 weeks before starting study treatment. Any symptoms attributed to brain metastases must be stable for at least 4 weeks before starting study treatment; radiographic stability should be determined by comparing contrast-enhanced computed tomography (CT) or magnetic resonance imaging (MRI) brain scan performed during screening to a prior scan performed at least 4 weeks earlier
10. Meningeal carcinomatosis
11. Significant cardiovascular impairment (history of congestive heart failure greater than New York Heart Association [NYHA] grade II, unstable angina or myocardial infarction within the past 6 months, or serious cardiac arrhythmia)
12. Electrocardiogram (ECG) with QT interval corrected for heart rate (QTc) interval greater than 470 msec (as measured either by Bazett's or Fredericia's formula)
13. Pre-existing neuropathy greater than Grade 2
14. Anti-coagulant therapy with warfarin or related compounds, other than for line patency, that cannot be changed to heparin-based therapy for the duration of the study
15. Subjects with known positive serology for Human Immunodeficiency Virus (HIV), or Hepatitis B or C
16. Subjects with other significant disease or disorder that, in the Investigator's opinion, would exclude the subject from the study
17. Major surgery within 4 weeks before starting study treatment or scheduled for surgery during the projected course of the study
18. Unable to swallow tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-01-26 (Actual); Primary Completion 2014-07-28 (Actual); Study Completion 2015-10-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Bulgaria (3):
  - Pleven
  - Plovdiv
  - Sofia
- Russia (4):
  - Chelyabinsk
  - Krasnodarsky Region
  - Saint Petersburg
  - Stavropol Krai
- United Kingdom (3):
  - Glasgow
  - Leeds
  - Newcastle upon Tyne

REFERENCES:
- [Derived] Twelves C, Anthoney A, Savulsky CI, Guo M, Reyderman L, Cresti N, Semiglazov V, Timcheva C, Zubairi I, Morrison R, Plummer R, Evans TRJ. A phase 1b/2, open-label, dose-escalation, and dose-confirmation study of eribulin mesilate in combination with capecitabine. Br J Cancer. 2019 Mar;120(6):579-586. doi: 10.1038/s41416-018-0366-5. Epub 2019 Feb 20. PMID 30783204

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 13 investigative sites in Bulgaria, Russia, and United Kingdom from 26 January 2010 to 13 October 2015.
Pre-assignment Details: Phase 1b (Dose Escalation Phase): total 43 participants with solid tumors were screened, of which 9 were screen failures and 34 received study treatment; Phase 2 (Dose Confirmation Phase): total 54 female participants with breast cancer were screened, of which 12 were screen failures and 42 received study treatment.
Groups:
- Phase 1b (Schedule 1): Eribulin Mesilate (1.2 mg/m^2): Participants received eribulin mesilate 1.2 milligrams per square meter (mg/m^2), injection, intravenously, once, on Day 1 and capecitabine 1000 mg/m^2, tablets, orally, twice daily from Day 1 to 14 in each 21-day treatment cycle for as long as the treatment was clinically appropriate according to the judgment of the investigator or until the occurrence of progressive disease (PD), undue toxicity, the presence of other medical conditions that prohibit continuation of therapy, pregnancy, a delay of more than 14 days in starting the next cycle during Phase 1b (Schedule 1).
- Phase 1b (Schedule 1): Eribulin Mesilate (1.6 mg/m^2): Participants received eribulin mesilate 1.6 mg/m^2, injection, intravenously, once, on Day 1 and capecitabine 1000 mg/m^2, tablets, orally, twice daily from Day 1 to 14 in each 21-day treatment cycle for as long as the treatment was clinically appropriate according to the judgment of the investigator or until the occurrence of PD, undue toxicity, the presence of other medical conditions that prohibit continuation of therapy, pregnancy, a delay of more than 14 days in starting the next cycle during Phase 1b (Schedule 1).
- Phase 1b (Schedule 1): Eribulin Mesilate (2.0 mg/m^2): Participants received eribulin mesilate 2.0 mg/m^2, injection, intravenously, once, on Day 1 and capecitabine 1000 mg/m^2, tablets, orally, twice daily from Day 1 to 14 in each 21-day treatment cycle for as long as the treatment was clinically appropriate according to the judgment of the investigator or until the occurrence of PD, undue toxicity, the presence of other medical conditions that prohibit continuation of therapy, pregnancy, a delay of more than 14 days in starting the next cycle during Phase 1b (Schedule 1).
- Phase 1b (Schedule 2): Eribulin Mesilate (0.7 mg/m^2): Participants received eribulin mesilate 0.7 mg/m^2, injection, intravenously, once, on Days 1 and 8, and capecitabine 1000 mg/m^2, tablets, orally, twice daily from Day 1 to 14 in each 21-day treatment cycle for as long as the treatment was clinically appropriate according to the judgment of the investigator or until the occurrence of PD, undue toxicity, the presence of other medical conditions that prohibit continuation of therapy, pregnancy, a delay of more than 14 days in starting the next cycle during Phase 1b (Schedule 2).
- Phase 1b (Schedule 2): Eribulin Mesilate (1.1 mg/m^2): Participants received eribulin mesilate 1.1 mg/m^2, injection, intravenously, once, on Days 1 and 8, and capecitabine 1000 mg/m^2, tablets, orally, twice daily from Day 1 to 14 in each 21-day treatment cycle for as long as the treatment was clinically appropriate according to the judgment of the investigator or until the occurrence of PD, undue toxicity, the presence of other medical conditions that prohibit continuation of therapy, pregnancy, a delay of more than 14 days in starting the next cycle during Phase 1b (Schedule 2).
- Phase 1b (Schedule 2): Eribulin Mesilate (1.4 mg/m^2): Participants received eribulin mesilate 1.4 mg/m^2, injection, intravenously, once, on Days 1 and 8, and capecitabine 1000 mg/m^2, tablets, orally, twice daily from Day 1 to 14 in each 21-day treatment cycle for as long as the treatment was clinically appropriate according to the judgment of the investigator or until the occurrence of PD, undue toxicity, the presence of other medical conditions that prohibit continuation of therapy, pregnancy, a delay of more than 14 days in starting the next cycle during Phase 1b (Schedule 2).
- Phase 2: Eribulin Mesilate 1.4 mg/m^2: Participants received eribulin mesilate 1.4 mg/m^2, injection, intravenously, once, on Days 1 and 8, and capecitabine 1000 mg/m^2, tablets, orally, twice daily from Day 1 to 14 in each 21-day treatment cycle for as long as the treatment was clinically appropriate according to the judgment of the investigator or until the occurrence of PD, undue toxicity, the presence of other medical conditions that prohibit continuation of therapy, pregnancy, a delay of more than 14 days in starting the next cycle during Phase 2.
Period: Phase 1b (Dose Escalation Phase)
Arm/Group | Phase 1b (Schedule 1): Eribulin Mesilate (1.2 mg/m^2) | Phase 1b (Schedule 1): Eribulin Mesilate (1.6 mg/m^2) | Phase 1b (Schedule 1): Eribulin Mesilate (2.0 mg/m^2) | Phase 1b (Schedule 2): Eribulin Mesilate (0.7 mg/m^2) | Phase 1b (Schedule 2): Eribulin Mesilate (1.1 mg/m^2) | Phase 1b (Schedule 2): Eribulin Mesilate (1.4 mg/m^2) | Phase 2: Eribulin Mesilate 1.4 mg/m^2
Started | 8 | 6 | 5 | 3 | 6 | 6 | 0
Completed | 5 | 4 | 4 | 3 | 3 | 3 | 0
Not Completed | 3 | 2 | 1 | 0 | 3 | 3 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 2 | 0 | 0
Not completed — Clinical Progression | 0 | 1 | 0 | 0 | 1 | 1 | 0
Period: Phase 2 (Dose-confirmation Phase)
Arm/Group | Phase 1b (Schedule 1): Eribulin Mesilate (1.2 mg/m^2) | Phase 1b (Schedule 1): Eribulin Mesilate (1.6 mg/m^2) | Phase 1b (Schedule 1): Eribulin Mesilate (2.0 mg/m^2) | Phase 1b (Schedule 2): Eribulin Mesilate (0.7 mg/m^2) | Phase 1b (Schedule 2): Eribulin Mesilate (1.1 mg/m^2) | Phase 1b (Schedule 2): Eribulin Mesilate (1.4 mg/m^2) | Phase 2: Eribulin Mesilate 1.4 mg/m^2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 42
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 25
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 17
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Clinical progression | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 8
Not completed — Investigators decision | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Development of bladder cancer | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Phase 1b (Schedule 1): Eribulin Mesilate (1.2 mg/m^2): Participants received eribulin mesilate 1.2 mg/m^2, injection, intravenously, once, on Day 1 and capecitabine 1000 mg/m^2, tablets, orally, twice daily from Day 1 to 14 in each 21-day treatment cycle for as long as the treatment was clinically appropriate according to the judgment of the investigator or until the occurrence of PD, undue toxicity, the presence of other medical conditions that prohibit continuation of therapy, pregnancy, a delay of more than 14 days in starting the next cycle during Phase 1b (Schedule 1).
- Total: Total of all reporting groups
Arm/Group | Phase 1b (Schedule 1): Eribulin Mesilate (1.2 mg/m^2) | Phase 1b (Schedule 1): Eribulin Mesilate (1.6 mg/m^2) | Phase 1b (Schedule 1): Eribulin Mesilate (2.0 mg/m^2) | Phase 1b (Schedule 2): Eribulin Mesilate (0.7 mg/m^2) | Phase 1b (Schedule 2): Eribulin Mesilate (1.1 mg/m^2) | Phase 1b (Schedule 2): Eribulin Mesilate (1.4 mg/m^2) | Phase 2: Eribulin Mesilate 1.4 mg/m^2 | Total
Number analyzed (Participants) | 8 | 6 | 5 | 3 | 6 | 6 | 42 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 3 | 2 | 5 | 3 | 37 | 61
  >=65 years | 1 | 2 | 2 | 1 | 1 | 3 | 5 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 3 | 2 | 3 | 5 | 42 | 61
  Male | 2 | 6 | 2 | 1 | 3 | 1 | 0 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 6 | 5 | 3 | 6 | 6 | 42 | 76
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 8 | 6 | 5 | 3 | 6 | 6 | 41 | 75
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose-limiting Toxicities (DLTs) as Per National Cancer Institute Common Terminology Criteria for Adverse Events Version 3.0 (NCI CTCAE v3.0)
Description: DLTs as per NCI CTCAE v3.0 were defined as:1) Neutropenia Grade 4 that lasted at least 7 days, 2) Neutropenia Grade 3 or 4 complicated by fever and/or infection (absolute neutrophil count [ANC] less than 1.0*10^9/liter [L], fever of at least 38.5 degree celsius [°C]), 3)Thrombocytopenia Grade 4, 4) Thrombocytopenia Grade 3 complicated by bleeding and/or requiring platelet or blood transfusion, 5) Non-hematological toxicity Grade 3 or higher (excluding Grade 3 nausea, and Grade 3 or 4 vomiting or diarrhea in participants who had not received optimal treatment with antiemetic and/or antidiarrheal medication; excluding laboratory abnormalities without clinical symptoms), 6) Delayed recovery from treatment-related toxicity resulting in dose delay greater than 14 days, 7) Failure to administer at least 75 percent (%) of planned study drugs during Cycle 1 as result of Grade 2 or higher treatment-related toxicity that constituted increase of at least 2 grades from baseline.
Time Frame: Cycle 1 (21 days)
Population: The safety set included the group of participants who received study drug and had at least 1 post dose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b (Schedule 1): Eribulin Mesilate (1.2 mg/m^2) | Phase 1b (Schedule 1): Eribulin Mesilate (1.6 mg/m^2) | Phase 1b (Schedule 1): Eribulin Mesilate (2.0 mg/m^2) | Phase 1b (Schedule 2): Eribulin Mesilate (0.7 mg/m^2) | Phase 1b (Schedule 2): Eribulin Mesilate (1.1 mg/m^2) | Phase 1b (Schedule 2): Eribulin Mesilate (1.4 mg/m^2)
Number analyzed (Participants) | 8 | 6 | 5 | 3 | 6 | 6
Participants | 1 | 1 | 2 | 0 | 1 | 1

2. Primary Outcome: Phase 2: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had either a confirmed complete response (CR) or partial response (PR). ORR was assessed based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v 1.1). CR was defined as disappearance of all target lesions. All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to less than (<) 10 millimeter (mm). PR was defined as at least a 30 percent (%) decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of the longest diameter. ORR was summarized using the Clopper-Pearson method.
Time Frame: From the first dose of study drug until PD or up to 30 days after the last dose of study treatment (up to approximately 3.75 years)
Population: The Dose-confirmation full analysis set included all participants who enrolled in the Dose-confirmation Cohort (Phase 2) and received at least 1 dose of drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Eribulin Mesilate 1.4 mg/m^2
Number analyzed (Participants) | 42
percentage of participants | 42.9 [27.7 to 59.0]

3. Secondary Outcome: Phase 2: Time to Response
Description: Time to response (CR or PR) was defined as the time from the first dose until first documented evidence of CR or PR (whichever status was recorded first). Time to response was assessed based on RECIST v 1.1. CR was defined as disappearance of all target lesions. All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to less than 10 mm. PR was defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of the longest diameter. Time to response was summarized using the Kaplan-Meier method.
Time Frame: From the first dose of study drug treatment start date until date of first documented evidence of CR or PR or up to 30 days after the last dose of study treatment (up to approximately 3.75 years)
Population: The Dose-confirmation full analysis set included all participants who enrolled in the Dose-confirmation Cohort (Phase 2) and received at least 1 dose of drug. Here "overall number of participants analyzed" signifies participants who had CR or PR.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2: Eribulin Mesilate 1.4 mg/m^2
Number analyzed (Participants) | 18
days | 44.0 [42.0 to 84.0]

4. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: DOR: time from first documented evidence of CR or PR until first documented sign of PD or death. DOR was assessed based on RECIST v 1.1. CR: disappearance of all target lesions. All pathological lymph nodes (whether target/non-target) must have a reduction in their short axis to >10 mm. PR: at least a 30% decrease in sum of longest diameter of target lesions, taking as reference the baseline sum of longest diameter. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study (this includes baseline sum if that is the smallest on study). DOR was summarized using the Kaplan-Meier method.
Time Frame: From date of the first CR or PR until the date of first documentation of PD or death or up to 30 days after the last dose of study treatment (up to approximately 3.75 years)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2: Eribulin Mesilate 1.4 mg/m^2
Number analyzed (Participants) | 18
days | 261.0 [161.0 to NA] — Here, NA means that the upper limit of 95% confidence interval (CI) was not estimable due to an insufficient number of events.

5. Secondary Outcome: Phase 2: Stable Disease (SD) Rate
Description: SD rate was defined as the percentage of participants with a SD that lasted for a minimum of 5 weeks. SD rate was assessed based on RECIST version 1.1. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PR: at least a 30% decrease in sum of longest diameter of target lesions, taking as reference the baseline sum of longest diameter. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study (this includes baseline sum if that is the smallest on study).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Eribulin Mesilate 1.4 mg/m^2
Number analyzed (Participants) | 42
percentage of participants | 38.1

6. Secondary Outcome: Phase 1b and Phase 2: Percentage of Participants With Non-CR/Non-PD
Description: Non-CR/Non-PD was for participants who had non-target disease only (minimum duration from randomization to Non-CR/Non-PD >=7 weeks) and assessed by investigator based on RECIST v1.1. Non-CR/Non-PD: persistence of one or more non-target lesions, maintenance of tumor marker level above the normal limits.
Time Frame: as for outcome 2
Population: Full Analysis Set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1b (Schedule 1): Eribulin Mesilate (1.2 mg/m^2) | Phase 1b (Schedule 1): Eribulin Mesilate (1.6 mg/m^2) | Phase 1b (Schedule 1): Eribulin Mesilate (2.0 mg/m^2) | Phase 1b (Schedule 2): Eribulin Mesilate (0.7 mg/m^2) | Phase 1b (Schedule 2): Eribulin Mesilate (1.1 mg/m^2) | Phase 1b (Schedule 2): Eribulin Mesilate (1.4 mg/m^2) | Phase 2: Eribulin Mesilate 1.4 mg/m^2
Number analyzed (Participants) | 8 | 6 | 5 | 3 | 6 | 6 | 42
percentage of participants | 0 | 0 | 0 | 0 | 16.7 | 0 | 0

7. Secondary Outcome: Phase 2: Duration of Stable Disease (SD)
Description: Duration of SD was measured from date of the first dose until progression. Duration of SD was assessed based on RECIST v1.1. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PR: at least a 30% decrease in sum of longest diameter of target lesions, taking as reference the baseline sum of longest diameter. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study (this includes baseline sum if that is the smallest on study). Duration of SD was summarized using the Kaplan-Meier method.
Time Frame: From the first dose of study drug until PD or 30 days after the last dose of study treatment (up to approximately 3.75 years)
Population: The Dose-confirmation full analysis set included all participants who enrolled in the Dose-confirmation Cohort (Phase 2) and received at least 1 dose of drug. Here "overall number of participants analyzed" signifies participants who had SD.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2: Eribulin Mesilate 1.4 mg/m^2
Number analyzed (Participants) | 16
days | 162.0 [91.0 to 330.0]

8. Secondary Outcome: Phase 2: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with a confirmed CR, PR, or SD divided by the number of participants in the analysis set. DCR was assessed by an investigator based on RECIST v1.1. CR: disappearance of all target lesions. All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to <10 mm. PR: at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of the longest diameter. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study (this includes baseline sum if that is the smallest on study). DCR was summarized using the Clopper-Pearson method.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Eribulin Mesilate 1.4 mg/m^2
Number analyzed (Participants) | 42
percentage of participants | 81.0 [65.9 to 91.4]

9. Secondary Outcome: Phase 2: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants with a confirmed CR, PR, or SD of at least 6 months duration (durable SD) divided by the number of participants in the analysis set. CBR was determined by an investigator based on RECIST v1.1. CR: disappearance of all target lesions. All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to <10 mm. PR: at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of the longest diameter. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study (this includes baseline sum if that is the smallest on study). CBR was summarized using the Clopper-Pearson method.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Eribulin Mesilate 1.4 mg/m^2
Number analyzed (Participants) | 42
percentage of participants | 57.1 [41.0 to 72.3]

10. Secondary Outcome: Phase 2: Progression-free Survival (PFS)
Description: PFS was defined as the time from the first dose date until PD or death due to any cause. PFS was determined by an investigator based on RECIST v1.1. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study (this includes baseline sum if that is the smallest on study). PFS was summarized using the Kaplan-Meier method.
Time Frame: From the first dose of study drug until PD or death due to any cause or 30 days after the last dose of study treatment (up to approximately 3.75 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2: Eribulin Mesilate 1.4 mg/m^2
Number analyzed (Participants) | 42
days | 219.0 [138.0 to 330.0]

ADVERSE EVENTS:
Time Frame: From date of first dose up to 30 days after the last dose of study treatment (up to approximately 3.75 years)
Description: The safety set included the group of participants who received study drug and had at least 1 post dose safety assessment.
Arm/Group | Phase 1b (Schedule 1): Eribulin Mesilate (1.2 mg/m^2) | Phase 1b (Schedule 1): Eribulin Mesilate (1.6 mg/m^2) | Phase 1b (Schedule 1): Eribulin Mesilate (2.0 mg/m^2) | Phase 1b (Schedule 2): Eribulin Mesilate (0.7 mg/m^2) | Phase 1b (Schedule 2): Eribulin Mesilate (1.1 mg/m^2) | Phase 1b (Schedule 2): Eribulin Mesilate (1.4 mg/m^2) | Phase 2: Eribulin Mesilate 1.4 mg/m^2
All-Cause Mortality (participants affected / at risk) | 1/8 | 1/6 | 0/5 | 0/3 | 1/6 | 2/6 | 3/42
Serious Adverse Events (participants affected / at risk) | 2/8 | 4/6 | 1/5 | 2/3 | 3/6 | 4/6 | 10/42
Other Adverse Events (participants affected / at risk) | 7/8 | 6/6 | 5/5 | 3/3 | 6/6 | 6/6 | 39/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b (Schedule 1): Eribulin Mesilate (1.2 mg/m^2) (N=8) | Phase 1b (Schedule 1): Eribulin Mesilate (1.6 mg/m^2) (N=6) | Phase 1b (Schedule 1): Eribulin Mesilate (2.0 mg/m^2) (N=5) | Phase 1b (Schedule 2): Eribulin Mesilate (0.7 mg/m^2) (N=3) | Phase 1b (Schedule 2): Eribulin Mesilate (1.1 mg/m^2) (N=6) | Phase 1b (Schedule 2): Eribulin Mesilate (1.4 mg/m^2) (N=6) | Phase 2: Eribulin Mesilate 1.4 mg/m^2 (N=42)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heparin-induced Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (4)
Device related infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant Ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal Cord Compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal Ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolongation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestine obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b (Schedule 1): Eribulin Mesilate (1.2 mg/m^2) (N=8) | Phase 1b (Schedule 1): Eribulin Mesilate (1.6 mg/m^2) (N=6) | Phase 1b (Schedule 1): Eribulin Mesilate (2.0 mg/m^2) (N=5) | Phase 1b (Schedule 2): Eribulin Mesilate (0.7 mg/m^2) (N=3) | Phase 1b (Schedule 2): Eribulin Mesilate (1.1 mg/m^2) (N=6) | Phase 1b (Schedule 2): Eribulin Mesilate (1.4 mg/m^2) (N=6) | Phase 2: Eribulin Mesilate 1.4 mg/m^2 (N=42)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (4) | 0 (0) | 0 (0) | 2 (3) | 5 (19) | 34 (238)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 20 (73)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 12 (24)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Nausea (Gastrointestinal disorders) | 4 (5) | 4 (9) | 4 (6) | 2 (4) | 3 (15) | 6 (24) | 12 (28)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 3 (3) | 1 (5) | 2 (6) | 3 (6) | 4 (13) | 8 (30)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 3 (6) | 0 (0) | 0 (0) | 2 (3) | 4 (6) | 8 (35)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 6 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (5) | 3 (6) | 0 (0) | 3 (7) | 6 (18) | 6 (9)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (3) | 1 (3) | 0 (0) | 2 (3) | 4 (6)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 1 (3) | 1 (2) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 2 (3) | 15 (26)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (5) | 0 (0) | 0 (0) | 1 (11) | 0 (0) | 11 (19)
Lethargy (Nervous system disorders) | 2 (3) | 4 (7) | 2 (4) | 2 (5) | 4 (22) | 4 (15) | 8 (66)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 8 (21)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (7)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 1 (1) | 6 (16)
Fatigue (General disorders) | 1 (2) | 1 (1) | 2 (7) | 0 (0) | 1 (1) | 2 (3) | 6 (10)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (15)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (9)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (7)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 5 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 4 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (6) | 1 (2) | 1 (2) | 3 (3) | 3 (6)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (4)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (11) | 1 (1) | 1 (3)
Paraesthesia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parasomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (3) | 2 (2) | 1 (3) | 2 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Plantar Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes